CLINICAL TRIAL: NCT04147299
Title: Cardiopulmonary and Right Ventricular Function in Health and Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 19-1141
Record Dates: First submitted 2019-10-02; First posted 2019-11-01 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Heart Failure; Athletes Heart
Keywords: Right Ventricular Function
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HFrEF: Heart Failure with Reduced Ejection Fraction
- HFpEF: Heart Failure with Preserved Ejection Fraction
- Elite Athletes: Endurance athletes

SUMMARY:
The primary objective of this research protocol is to advance the understanding of cardiopulmonary and right ventricular (RV) performance among individuals with cardiomyopathy (heart failure with reduced ejection fraction [HFrEF], heart failure with preserved ejection fraction [HFpEF]), as well as athletes engaging in endurance/prolonged exercise, who are at a high risk of an acquired cardiomyopathy during/following completion of an endurance event.

DETAILED DESCRIPTION:
For completion of specific aims 1-2, the protocol will be identical. Specific aim 1 involves analysis of patients with HFrEF as defined above; specific aim 2 involves analysis of patients with HFpEF as defined above. The protocol for specific aim 3 (analysis of endurance athletes) incorporates a different protocol than that described for specific aims 1-2.

For HFrEF and HFpEF patients (specific aims 1-2): There will be a single visit for testing. This visit will involve a baseline assessment of hemodynamics using a Swan-Ganz catheter, followed by invasive exercise testing with a high-fidelity conductance catheter, which provides the real-time RV PV loops. The Swan-Ganz catheter is a 7-French flexible catheter that is routinely used for hemodynamic assessment for clinical and research purposes (we are currently using this catheter for COMIRB #16-1635, and COMIRB #17-1042). The purpose of this catheter is to determine baseline hemodynamic parameters (in "layman's terms", to describe left and right-sided filling pressures, as well as pressures in the lungs), and to determine resting cardiac output. The Swan-Ganz catheter will be inserted and removed after obtaining these measurements - it is anticipated that this procedure will take 10-15 minutes. The primary investigator for this study, Dr. Cornwell, routinely performs these procedures in both clinical and research settings, and will use standard techniques for catheter insertion. Ultrasound guidance will be used to identify the right internal jugular vein, where the catheter is inserted, and fluoroscopy will be used to guide placement of the catheter for hemodynamic monitoring.

After completion of the baseline hemodynamic assessment, the Swan-Ganz catheter will be removed. Thereafter, the high-fidelity conductance catheter will be inserted into the RV using standard techniques. This catheter is also a 7-French flexible catheter (currently being used for COMIRB #17-1042) that has a pressure manometer on the tip, along with several conductance electrodes that continuously measure volume in the ventricle - by continuously recording changes in pressure and volume throughout the cardiac cycle, the catheter generates the "PV loop". These catheters provide information that is not available with standard Swan-Ganz catheters (refer to outcome measures listed above). Following insertion of the conductance catheter, an arterial line will be placed in either the left or right radial artery, using sterile technique and with ultrasound-guidance. The purpose of this catheter is two-fold: 1) to provide a gold-standard assessment of BP during exercise; and 2) to measure arterial oxygen saturation to calculate a cardiac output from the Fick equation. Baseline hemodynamic assessment will involve monitoring for approximately 5 minutes during spontaneous breathing, followed by approximately 6 minutes of breathing at a controlled respiratory rate (12 times per minute), which allows for determination of short-term blood pressure variability after controlling for the effect of respiratory variation, followed by Valsalva maneuver and vasomotor reactivity (inspiratory breath-hold for 30 seconds).

Following insertion of the conductance catheter, arterial catheter and acquisition of baseline data, the patient will be positioned on an upright cycle ergometer. In the event that the patient is not able to perform upright exercise, a supine ergometer will be used. The patient will then complete exercise at two submaximal workloads (below their ventilatory threshold) that simulate real-world scenarios/normal activities of daily living, followed by peak exercise. To obtain submaximal data, workload on the bicycle will begin at 0 Watts. Every 1-2 minutes, workload will be steadily increased, generally in 12.5-25 Watt-increments, until the patient indicates that the rate-of-perceived exertion (RPE) score is 7-9, on a 6-20 point scale.24 This workload will correspond to "mild" exercise, or steady-state 1. Workload will be held at this level for approximately 4-5 minutes, during which time hemodynamic data will be obtained. Thereafter, workload will again be increased in 12.5-25 Watt increments until the participate indicates that the RPE score is 11-13.24 This workload will correspond to a "moderate" exercise, or steady-state 2. Workload will be held at this level for approximately 4-5 minutes, during which time hemodynamic data will be obtained. The patient will then be allotted a 5-10 minute break. After the break, the patient will complete a symptom-limited cardiopulmonary exercise test, whereby workload will begin at 0 Watts, and generally increase every 1-2 minutes in 12.5-25 Watt increments until exhaustion. Hemodynamic data will be continuously recorded, and final data will be obtained at the peak workload achieved. This protocol will allow for acquisition of data at five different positions: 1) supine rest; 2) upright rest; 3) steady-state 1, or "mild" exercise; 4) steady-state 2, or "moderate" exercise; and 5) peak exercise. Blood samples will be collected at each of these stages: blood will be tested for arterial and venous oxygen saturation levels (to calculate a Fick cardiac output), as well as a venous/capillary lactic acid level by finger stick. Lactic acid levels will be used to assess the participant's work effort at each stage of exercise (as a "rule-of-thumb", submaximal levels of exercise have an associated lactic acid level of below 4mmol/L. A complete blood count will be obtained in the supine resting position to determine hemoglobin concentration, which will be used to calculate Fick cardiac output during all stages of exercise. Following completion of the study, the patient will be returned to a supine position and de-instrumented. This protocol is very similar to protocols used as part of COMIRB #16-1635 and #17-1042; based on our experience with these protocols, it is anticipated that this study will last approximately 4-5 hours.

For Endurance Athletes (specific aim 3): There will be two visits for this study:

* Visit 1: Baseline Assessment: this visit will include informed consent, study enrollment, history and physical, followed by a non-invasive cardiopulmonary exercise test (CPET) with stress echocardiography. The CPET will be conducted in the following manner: a resting echocardiogram will be performed to assess cardiac structure and function and rule-out any structural disease. The athlete will then complete a symptom-limited CPET, whereby workload on the ergometer will start at 0 Watts, and increase by approximately 50-Watt increments every 1-2 minutes until exhaustion. Immediately following completion of the test, echocardiography will be repeated to assess wall motion and cardiac structure at peak exercise. During this test, heart rate (HR) and rhythm, as well as blood pressure (BP) will be continuously monitored non-invasively. In the event that any abnormalities are detected during this period of time, the patient will be excluded from further testing. Results of the test will be communicated with the participant.
* Visit 2: "Race-Day". On this day of testing, participants will complete a non-contrast cardiac MRI prior to and immediately following testing. Testing will include a timed-trial for completion of a 180km cycling event (the distance of the bicycling portion of an Ironman event)22.

  * Baseline cardiac MRI: to evaluate baseline cardiac structure and function. This will be completed in the Brain Imaging Center at the Anschutz Medical Campus.
  * Testing: after completion of cardiac MRI, participants will be escorted to laboratory for testing. Athletes will undergo insertion of a Swan-Ganz catheter using standard techniques (as described above). Baseline hemodynamic assessment will be obtained to determine left and right-sided filling pressures, as well as cardiac output. Spontaneous and controlled breathing, as well as Valsalva maneuver and vasomotor reactivity, will also be obtained. Following this assessment, the Swan-Ganz catheter will be removed and a conductance catheter will be inserted in order to obtain RV PV loops. Supine resting loops will be acquired. Thereafter, the athlete will be positioned on an upright bicycle. The participant will then complete a timed-trial (ie, we will record the time required to completion of the event). The distance will be the same for all participants and will be 180km (the distance of the cycling portion of an Ironman competition)22. Participants will be instructed to complete the event at a pace that they are comfortable with and is compatible with their typical racing pace. Breaks during cycling will be allotted at the athlete's request. Food and drink/snacks will be allotted at the athlete's request (the goal is to simulate a real-world race-day scenario). During the event, HR and rhythm, as well as BP, will be continuously recorded. RV PV loops, as well as gas-exchange metrics via indirect calorimetry, will be analyzed continuously and recorded every 30 minutes during the event. Following completion of the event, the athlete will be placed back in supine position, and post-event hemodynamic assessment will be completed. This will include acquisition of resting RV PV loops from the conductance catheter, followed by re-insertion of the Swan-Ganz catheter for spontaneous and controlled breathing, as well as a Valsalva maneuver and vasomotor reactivity. The participant will then be de-instrumented and the test-phase completed. Based on our experience with performing similar assessments, coupled with typical cycling times to complete 180km cycling events, it is anticipated that this test will take ~6 hours to complete.
  * Post-Test cardiac MRI: to evaluate cardiac structure and function following completion of test.

ELIGIBILITY:
Heart failure with reduced ejection fraction (HFrEF):

1. Inclusion criteria:

   1. Individuals with clinical heart failure, with left ventricular ejection fraction < 50% on a recent echocardiogram within past 6 months.
   2. Patients must be ambulatory, clinically stable and able to perform exercise on a stationary bicycle.
   3. Preserved right ventricular function. Right ventricular dysfunction will be defined by: imaging evidence of RV dysfunction on echocardiogram, with tricuspid annular plane systolic excursion (TAPSE) < 17mm6; hemodynamic evidence of RV dysfunction, defined by elevated right-sided filling pressures (RAP) on a clinically obtained right heart catheterization and a ratio of RAP to pulmonary capillary wedge ratio (PCWP) greater than two-thirds; clinical evidence of RV dysfunction, defined by elevated jugular venous pulsations and 3-4+ peripheral edema.
2. Exclusion criteria:

   1. Non-cardiac factors that preclude the ability to exercise, such as (but not limited to) osteoarthritis or any other musculoskeletal disease; peripheral vascular disease.
   2. Uncontrolled atrial or ventricular arrhythmias
   3. Significant valvular disease (>mild stenosis, >moderate regurgitation), cor pulmonale, significant pulmonary disease, congenital heart disease, left-to-right shunt, unstable coronary artery disease, hypertrophic cardiomyopathy, high-output heart failure, or constrictive pericarditis.
   4. The primary-investigator will reserve authority to use best clinical judgment to exclude patients from consideration for participation as case-based situations arise.
   5. Any acute/recent illness that would render the individual unable to participate in this study, as determined by the primary investigator.

Heart failure with preserved ejection fraction (HFpEF):

1. Inclusion criteria:

   1. individuals with clinical heart failure symptoms, but with left ventricular ejection fraction 50% or greater on a recent echocardiogram within past 6 months. Patients must have imaging evidence of diastolic dysfunction, such as an E/e' ratio > 14, evidence of grade 2 or greater diastolic dysfunction or a restrictive filling pattern on imaging.
   2. Patients must have an elevated brain-natriuretic peptide (BNP) of 80+ pg/ml (ever) or an NT-pro BNP of 125+ pg/ml (ever). Patients must be ambulatory and able to perform exercise on a stationary bicycle.
   3. If patients have a normal BNP (or NT-pro BNP), they must have a history of elevated left-sided filling pressures (e.g. PCWP, or left ventricular end-diastolic pressure) > 15mmHg on a clinically-indicated right heart catheterization at rest, or 25+mmHg during exercise.
   4. Preserved right ventricular function. Right ventricular dysfunction will be defined by: imaging evidence of RV dysfunction on echocardiogram, with tricuspid annular plane systolic excursion (TAPSE) < 17mm6; hemodynamic evidence of RV dysfunction, defined by elevated right-sided filling pressures (RAP) on a clinically obtained right heart catheterization and a ratio of RAP to pulmonary capillary wedge ratio (PCWP) greater than two-thirds; clinical evidence of RV dysfunction, defined by elevated jugular venous pulsations and 3-4+ peripheral edema.
2. Exclusion criteria:

   1. Non-cardiac factors that preclude the ability to exercise, such as (but not limited to) osteoarthritis or any other musculoskeletal disease; peripheral vascular disease.
   2. Uncontrolled atrial or ventricular arrhythmias
   3. Significant valvular disease (>mild stenosis, >moderate regurgitation), cor pulmonale, significant pulmonary disease, congenital heart disease, left-to-right shunt, unstable coronary artery disease, hypertrophic cardiomyopathy, high-output heart failure, or constrictive pericarditis.
   4. The primary-investigator will reserve authority to use best clinical judgment to exclude patients from consideration for participation as case-based situations arise.
   5. Any acute/recent illness that would render the individual unable to participate in this study, as determined by the primary investigator.

Endurance athletes:

1. Inclusion criteria

   1. Individuals 18+ years of age who participate in endurance exercise primarily through bicycling (e.g. cyclists or triathletes)
   2. Individuals must spend approximately 8-10 hours per week on exercise training
   3. Compete regularly in competitive endurance/cycling events, and perform well, having finished a competition in top 25% of competitors
2. Exclusion criteria:

   1. Any known history of structural cardiovascular disease
   2. History of an adverse cardiovascular event during/immediately following a competition - e.g. syncope, cardiac arrest
   3. History of placement of an automatic implantable cardioverter-defibrillator
   4. Personal use of performance-enhancing drugs

Ages: 18 Years to 89 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: HFrEF - 20 participants - Individuals with clinical heart failure, with left ventricular ejection fraction < 50% on a recent echocardiogram within past 6 months.
  HFpEF - 20 participants - Individuals with clinical heart failure symptoms, but with left ventricular ejection fraction 50% or greater on a recent echocardiogram within past 6 months. Patients must have imaging evidence of diastolic dysfunction, such as an E/e' ratio > 14, evidence of grade 2 or greater diastolic dysfunction or a restrictive filling pattern on imaging.
  Elite/Endurance Athletes - 20 participants - Individuals 18+ years of age who participate in endurance exercise primarily through bicycling (e.g. cyclists or triathletes)
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-02-15 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Cardiac output | 1-2 years
  measured in L/min from the catheter during exercise.
Contractility | 1-2 years
  measured by dpdt, mmHg/sec
Diastolic function | 1-2 years
  measured by dpdt, mmHg/sec

CONTACTS AND LOCATIONS:
Overall Officials: William Cornwell, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to disclose individual data at this time.